CLINICAL TRIAL: NCT00218296
Title: Treatment of Smokeless Tobacco Users
Brief Title: Comparison Across Treatment Conditions to Reduce Smokeless Tobacco Use
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIDA-14404-4; R01-DA14404-4; DPMCDA; R01DA014404 (NIH)
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Results first posted 2013-12-19 (Estimated); Last update posted 2017-10-16 (Actual); Status verified 2017-09

CONDITIONS: Tobacco Use Disorder
Keywords: Nicotine Dependence; Tobacco Dependence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care Group (Active Comparator): Usual care for cessation with immediate quit date scheduled and two weeks of nicotine patch supplied.
  Interventions: Drug: Usual Care Group
- Reduction Group (Experimental): Reduction in nicotine exposure for 6 weeks prior to quit date using medicinal nicotine lozenge or reduced nicotine smokeless tobacco.
  Interventions: Other: Reduction Group

INTERVENTIONS:
Drug: Usual Care Group — Nicotine replacement therapy
  Other Names: 21 mg Nicotine Patch; Nicoderm
  Arms: Usual Care Group
Other: Reduction Group — Subject selects preferred method for reduction.
  Other Names: Commit Nicotine Lozenge or; Reduced nicotine smokeless tobacco products (Skoal, Skoal Bandits)
  Arms: Reduction Group

SUMMARY:
Smokeless tobacco (ST), which includes both chewing tobacco and snuff, has health risks associated with its use. While treatment programs that focus on stopping tobacco use may be effective, past research has shown that interventions that specifically focus on reducing tobacco use may be equally effective and may motivate individuals to eventually quit using tobacco. This study will compare the effectiveness of a ST reduction treatment program versus a usual tobacco cessation treatment program (immediate cessation) for reducing tobacco use in ST users.

DETAILED DESCRIPTION:
Individuals who use ST are at increased risk for cancer or dying from cardiovascular disease. Other long-term effects include tooth abrasion, gum recession, and loss of bone in the jaw. Many individuals who use ST recognize the health risks associated with ST, but either do not want to quit or feel that it is impossible to quit. For these individuals, tobacco reduction may be an important transitional goal, either prior to quitting or as a treatment endpoint. By participating in a tobacco reduction program, these individuals may be motivated to eventually stop using tobacco altogether. The purpose of this study is to compare a ST reduction treatment program versus a standard tobacco cessation treatment program (immediate cessation) for reducing tobacco use in ST users.

This study will enroll regular users of ST. Participants will be randomly assigned to either a tobacco reduction program or to usual care, a standard tobacco cessation program during the first telephone contact. At the first clinic visit, participants assigned to the tobacco Reduction Group will replace their usual brand of ST with one of two options: an ST brand with less nicotine or nicotine lozenge. Participants will be encouraged to reduce their nicotine intake by at least 50% the first two weeks and encouraged to further reduce their nicotine intake in the following 4 weeks. Participants assigned to the Usual Care Group will be advised to quit and will be asked to set a quit date within two weeks. Telephone counseling, ideas on methods for sustaining cessation, and a self-help manual will also be provided along with a 2 week supply of nicotine patches. Study visits will occur at 2, 4, 8, 12, 26, and 32 (for reduction group) weeks. Outcome assessments will include vital signs, physiological measures related to tobacco use, levels of nicotine reduction, tobacco use status, and measures of motivation and self-efficacy to quit.

ELIGIBILITY:
Inclusion Criteria:

* No interest in stopping ST use within 90 days of study entry
* Daily use of ST in the 6 months prior to study entry

Exclusion Criteria:

* Current use of tobacco or nicotine products, other than ST
* Current unstable medical and mental health conditions
* Use of any medication that may affect tobacco use or be affected by a reduction in tobacco use
* Pregnant or breastfeeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2006-11; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Hatsukami, PhD, Principal Investigator — University of Minnesota
Locations (1):
- Univerisity of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Result] Schiller KR, Luo X, Anderson AJ, Jensen JA, Allen SS, Hatsukami DK. Comparing an immediate cessation versus reduction approach to smokeless tobacco cessation. Nicotine Tob Res. 2012 Aug;14(8):902-9. doi: 10.1093/ntr/ntr302. Epub 2012 Jan 4. PMID 22218402
- See also: Schiller KR, Luo X, Anderson AJ, Jensen JA, Allen SS, Hatsukami DK. Comparing an immediate cessation versus reduction approach to smokeless tobacco cessation. Nicotine Tob Res 2012. — http://www.ncbi.nlm.nih.gov/pubmed/22218402

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 3/2007 through 5/2008.
Pre-assignment Details: Subjects who called the clinic were randomized to usual care (immediate cessation) or tobacco reduction to quit. Those who did not meet eligibility criteria at their first clinic visit due to unstable health, tobacco use rate, or other exclusionary criteria were dropped from the study.
Groups:
- Usual Care Group: Usual Care consisted of setting an immediate quit date and receiving 2 weeks of nicotine patch and behavioral counseling during the 6 week intervention period.
- Reduction Group: Subjects are instructed to reduce their tobacco use by 50% and then 75% over 6 weeks prior to quit date. Reduction is facilitated by using nicotine lozenge or ST brand switching resulting in reduced nicotine exposure.
Period: Overall Study
Arm/Group | Usual Care Group | Reduction Group
Started (Randomized at phone screen.) | 163 | 169
Attended Visti | 97 | 102
Completed | 52 | 48
Not Completed | 111 | 121
Not completed — Lost to Follow-up | 9 | 7
Not completed — Withdrawal by Subject | 36 | 47
Not completed — Randomized but did not enter treatment | 66 | 67

BASELINE CHARACTERISTICS:
Groups:
- Usual Care Group: Usual care consisted of setting an immediate quit date and receiving 2 weeks nicotine patch and behavioral counseling during the intervention period.
- Reduction Group: Subjects are instructed to reduce their tobacco use by 50% and then 75% over 6 weeks prior to quit date using nicotine lozenge or brand switching resulting in reduced nicotine exposure.
- Total: Total of all reporting groups
Arm/Group | Usual Care Group | Reduction Group | Total
Number analyzed (Participants) | 97 | 102 | 199
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 97 | 102 | 199
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.4 (8.4) | 35.1 (8.6) | 34.8 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 97 | 102 | 199
Region of Enrollment [Number; unit: participants]
  United States | 97 | 102 | 199

OUTCOME MEASURES:

1. Primary Outcome: Percent Abstinent From Tobacco at Week 12 (7 Day Point Prevalence)
Description: No tobacco use 7 days prior to Week 12 verified by biomarkers (urine, cotinine and CO)
Time Frame: 12 weeks
Population: Intent to treat
Measure: Number; unit: percentage of randomized
Arm/Group | Usual Care Group | Reduction Group
Number analyzed (Participants) | 163 | 169
percentage of randomized | 31 | 17
Statistical Analysis 1: Comparison: Usual Care Group vs Reduction Group; The null hypothesis was that the Usual Care Group (i.e. the immediate cessation group) and the Reduction Group had the same cessation rate. The alternative hypothesis was that they had different cessation rates. Two-sided test with a type I error of 0.05 was used; Test type: Superiority or Other; p = 0.04, Chi-squared; There were no adjustments in the analysis; Odds Ratio (OR) = 0.51, 95% CI 2-sided [0.26 to 0.99] — The reference group for the odds ratio estimate is the usual care condition, i.e., the immediate cessation condition

2. Primary Outcome: Percent Prolonged Abstinence From Tobacco at Week 12
Description: Continuous tobacco cessation from quit date through Week 12 verified by biomarkers (urine, cotinine and CO)
Time Frame: 12 weeks
Measure: Number; unit: percentage of randomized
Groups:
- Reduction Group: Reduction group subjects are instructed to reduce their tobacco use by 50% and then 75% over 6 weeks prior to quit date. Reduction is facilitated using nicotine lozenge or brand switching resulting in reduced nicotine exposure.
Arm/Group | Usual Care Group | Reduction Group
Number analyzed (Participants) | 163 | 169
percentage of randomized | 13 | 4
Statistical Analysis 1: Comparison: Usual Care Group vs Reduction Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.019, Chi-squared; There were no adjustments in the analysis; Odds Ratio (OR) = 0.28, 95% CI 2-sided [0.07 to 0.83] — The reference group for the odds ratio estimate is the Usual Care condition, i.e., the immediate cessation condition

3. Primary Outcome: Percent Abstinent From Tobacco at Week 26 (7 Day Point Prevalence)
Description: Abstinence from tobacco 7 days prior to Week 26 (Assessed at 26 weeks for Usual Care and 20 weeks for Reduction Group post-quit date)
Time Frame: 26 week
Measure: Number; unit: percentage of randomized
Arm/Group | Usual Care Group | Reduction Group
Number analyzed (Participants) | 163 | 169
percentage of randomized | 20 | 10
Statistical Analysis 1: Comparison: Usual Care Group vs Reduction Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.03, Chi-squared; There were no adjustments in the analysis; Odds Ratio (OR) = 0.42, 95% CI 2-sided [0.18 to 0.94] — The reference group for the odds ratio estimate is the usual care condition, i.e., the immediate cessation condition

4. Primary Outcome: Percent Prolonged Abstinence From Tobacco at Week 26
Description: Continuous Abstinence from quit date through Week 26 (Assessed at Week 26 for Usual Care and Week 20 for Reduction Group, Reduction Group's quit date is 6 weeks later than Usual Care).
Time Frame: 26 weeks
Population: Intent to treat
Measure: Number; unit: percentage of randomized
Arm/Group | Usual Care Group | Reduction Group
Number analyzed (Participants) | 163 | 169
percentage of randomized | 11 | 1
Statistical Analysis 1: Comparison: Usual Care Group vs Reduction Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = .002, Chi-squared; There were no adjustments in the analysis; Odds Ratio (OR) = 0.09, 95% CI 2-sided [0.004 to 0.48] — The reference group for the odds ratio estimate is the Usual Care Condition, i.e., the immediate cessation condition

5. Primary Outcome: Percent Abstinent From Tobacco at Week 32 (7 Day Point Prevalence)
Description: Abstinence from tobacco 7 days prior to Week 26 (Assessed at Week 32 for Usual Care and Week 26 for Reduction Group. Reduction Group's quit date is 6 weeks later than Usual Care).
Time Frame: 32 Weeks
Measure: Number; unit: percentage of randomized
Arm/Group | Usual Care Group | Reduction Group
Number analyzed (Participants) | 163 | 169
percentage of randomized | 20 | 11
Statistical Analysis 1: Comparison: Usual Care Group vs Reduction Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.056, Chi-squared; There were no adjustments in the analysis; Odds Ratio (OR) = 0.47, 95% CI 2-sided [0.20 to 1.03] — The reference group for the odds ratio estimate is the Usual Care Condition, i.e., the immediate cessation condition

6. Primary Outcome: Percent Prolonged Abstinence From Tobacco at Week 32
Description: Continuous Abstinence from quit date through Week 32 (Assessed at Week 32 for Usual Care and Week 26 for Reduction Group, Reduction Group's quit date is 6 weeks later than Usual Care).
Time Frame: 32 Weeks
Measure: Number; unit: percentage of randomized
Arm/Group | Usual Care Group | Reduction Group
Number analyzed (Participants) | 163 | 169
percentage of randomized | 11 | 1
Statistical Analysis 1: Comparison: Usual Care Group vs Reduction Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.002, Chi-squared — There were no adjustments in the analysis; Odds Ratio (OR) = 0.09, 95% CI 2-sided [0.004 to 0.48] — The reference group for the odds ratio estimate is the Usual Care Condition, i.e., the immediate cessation condition

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Usual Care Group | Reduction Group
Serious Adverse Events (participants affected / at risk) | 0/97 | 0/102
Other Adverse Events (participants affected / at risk) | 46/97 | 25/102
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care Group (N=97) | Reduction Group (N=102)
Sleep Disturbance (General disorders) | 19 (19) | 3 (3)
Dry Mouth (General disorders) | 4 (4) | 9 (12)
Headache (General disorders) | 8 (8) | 13 (18)
Muscle Aches (Musculoskeletal and connective tissue disorders) | 6 (7) | 0 (0)
Redness at Patch Site (General disorders) | 8 (8) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 21 (22) | 0 (0)

LIMITATIONS AND CAVEATS:
Sample size was limited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No